CLINICAL TRIAL: NCT05499208
Title: The Effect of Turning and Movement System on Breastfeeding Success, Pain and Comfort in Postpartum Cesarean Section
Brief Title: Rotation and Movement System, Postpartum Cesarean Sections
Acronym: Rotation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kars Harakani State Hospital (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Merve Lazoğlu, PhD student, Kars Harakani State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KarsHarakani Lazoglu0001
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Feeding, Exclusive
Keywords: pain; midwife; breast-feeding; movement; comfort
MeSH Terms: conditions — Breast Feeding; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giving side position with patient turning and movement system (Experimental): On the day she was admitted to the clinic, the pregnant woman was taken to the room with the turning and movement system, the system was introduced and the personal information form was filled. When she came to the clinic from the operating room, the puerperant was placed on the bed with the turning and motion system (side position) and a follow-up form for LATCH, GKO and Lactogenesis Free symptoms was filled in the first three breastfeedings. Before discharge, LATCH, GCS, and Lactogenesis symptoms follow-up forms were filled in the last three breastfeedings. WHO was filled 1-2 hours before discharge. On the 3rd and 4th days after discharge, the lactogenesis symptoms follow-up form was filled by phone.
  Interventions: Other: Giving side position with patient turning and movement system
- Control: Assigned Interventions standard care group (No Intervention): routine maintenance of the hospital

INTERVENTIONS:
Other: Giving side position with patient turning and movement system — To provide effective breastfeeding by placing the mother in position.
  Arms: Giving side position with patient turning and movement system

SUMMARY:
In the first half hour of a cesarean advertisement, the service-oriented mother will not be mobile and will need support to get fit in bed and start getting started. The patient turning and movement system will provide a lot of convenience to the mother who does not have enough support.

With the remote control system, the mother will be easily turned to the desired side in the bed and it will be ensured that she takes the desired position with less pain and more comfort.

DETAILED DESCRIPTION:
While studies on the Patient Turning and Movement System have been conducted on long-term bedridden patients, there is no scientific study examining its effects in the obstetric field. For the reasons mentioned above, the aim of this research is; The aim of this study is to investigate the effect of Patient Turning and Movement System on postpartum early postpartum breastfeeding success, pain and postpartum comfort in puerperant women who delivered by cesarean section and to contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35.
* Primiparity.
* Having a transverse cesarean section.
* At least primary school graduate.
* No high-risk pregnancy.
* Absence of any complications in the puerperal and newborn during the delivery and postnatal period

Exclusion Criteria:

* Having an open wound on the body and/or an allergic disease diagnosis on the skin.
* Development of puerperal complications (bleeding, infection, fever).
* At risk of convulsions; have diseases such as eclampsia, epilepsy.
* Having a body mass index above 40 (morbidly obese).
* Having any contraindications for breastfeeding.
* Having chronic opioid, antidepressant, and psychoactive drug use.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
The Effect of Turning and Movement System on Breastfeeding Success, Pain and Comfort in Postpartum Cesarean Section | two day
  It is a randomized study planned as a research. The sample of the study consists of postpartum women (75 experimental group, 75 control group) who had cesarean section. Breastfeeding success of postpartum women was evaluated with the LATCH Breastfeeding Diagnosis and Evaluation tool. This scale consists of five evaluation criteria (L:Latch on the brest, A: Audible Swallowing, T: Type of Nipple, C:Comfort of Breast/ Nipple, H: Hold/ Position). Each item is evaluated between 0-2 points. The scale has no breakpoints. The highest score that can be obtained from the scale is 10 and the lowest score is 0. An increase in the score obtained from the scale indicates the success of breastfeeding.
The Effect of Turning and Movement System on Breastfeeding Success, Pain and Comfort in Postpartum Cesarean Section | two days
  Postpartum pain was assessed with the Visual Comparison Scale. Painlessness on one head and the most severe pain on the other side were evaluated with a 10 cm ruler. An increase in the scale score indicates an increase in the severity of pain.

SECONDARY OUTCOMES:
The Effect of Turning and Movement System on Breastfeeding Success, Pain and Comfort in Postpartum Cesarean Section | one day
  Postpartum comfort of postpartum women was evaluated with the postpartum comfort scale. The scale has no breakpoints. The scale consists of 34 items. The minimum score to be taken from the scale is 34 and the maximum score is 170. The higher the score obtained from the scale, the higher the comfort.

CONTACTS AND LOCATIONS:
Overall Officials: merve lazoglu, phd, Principal Investigator — Kars Harakani State Hospital; Serap Ejder Apay, Prof., Study Director — Ataturk University Faculty of Health Sciences Department of Midwifery
Locations (1):
- Kars Harakani State Hospital, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
bireysel katılımcı verilerini diğer araştırmacılarla paylaşmıyoruz